CLINICAL TRIAL: NCT00564824
Title: The Impact of Caffeine on Brachial Endothelial Function in Healthy Subjects & in Patients With Ischemic Heart Disease
Brief Title: The Impact of Caffeine on Brachial Endothelial Function in Healthy Subjects and in Patients With Ischemic Heart Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Michael Shechter, MD, PI, Heart Institute, Sheba Medical Center
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: SHEBA-07-4913-MS-CTIL
Record Dates: First submitted 2007-11-27; First posted 2007-11-28 (Estimated); Last update posted 2010-02-25 (Estimated); Status verified 2010-02

CONDITIONS: Coronary Disease
Keywords: coronary disease; atherosclerosis; endothelial function; caffeine; cerebrovascular disease; prevention
MeSH Terms: conditions — Coronary Disease; Atherosclerosis; Cerebrovascular Disorders | interventions — Caffeine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- CAD patients (Experimental): Patients with prior history of coronary artery disease (CAD) (myocardial infarction, cerebrovascular accident, coronary angioplasty, S/p CABG operation) who will be given on the first day either caffeine of placebo tablet and 1-2 hours thereafter a brachial artery endothelial function testing (BRT) will be assessed for measuring the FMD. After 1 week the patients will come for a second BRT on placebo/caffeine tablets. If the patient received caffeine tablet the first BRT, he will be receiving placebo tablet the second week, however, if the patient received placebo the first BRT, a caffeine tablet will be given prior to the second BRT.
  Interventions: Drug: Caffeine
- Placebo (Experimental): Patients with prior history of coronary artery disease (CAD) (myocardial infarction, cerebrovascular accident, coronary angioplasty, S/p CABG operation) who will be given on the first day either caffeine of placebo tablet and 1-2 hours thereafter a brachial artery endothelial function testing (BRT) will be assessed for measuring the FMD. After 1 week the patients will come for a second BRT on placebo/caffeine tablets. If the patient received caffeine tablet the first BRT, he will be receiving placebo tablet the second week, however, if the patient received placebo the first BRT, a caffeine tablet will be given prior to the second BRT.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Caffeine — Caffeine 200 mg tablet
  Arms: CAD patients
Drug: Placebo — Placebo pills
  Arms: Placebo

SUMMARY:
Prior work (Chris, M. et al, Clinical Science 2005; 109, 55-60) has demonstrated that drinking a cup of coffee (80-100 mg of caffeine) an hour before endothelium-dependent FMD (flow-mediated dilatation) of the brachial artery, effects endothelial function in healthy adults subjects.

This effect might be attributed to caffeine, given that decaffeinated coffee (<2 mg of caffeine) was not associated with any change in endothelial performance.

In the current study we intend to further examine the impact of caffeine on brachial endothelial function among healthy subjects & in patients with proven ischemic heart disease.

DETAILED DESCRIPTION:
Background:

Prior work (Chris, M. et al, Clinical Science 2005; 109, 55-60) has demonstrated that drinking a cup of coffee (80-100 mg of caffeine) an hour before endothelium-dependent FMD (flow-mediated dilatation) of the brachial artery, effects endothelial function in healthy adults subjects.

This effect might be attributed to caffeine, given that decaffeinated coffee (<2 mg of caffeine) was not associated with any change in endothelial performance.

In the current study we intend to further examine the impact of caffeine on brachial endothelial function among healthy subjects & in patients with proven ischemic heart disease.

Aim:

To evaluate the impact of 200 mg caffeine tablet intake (equivalent to 2 cups of coffee), compared to placebo on brachial endothelial function in healthy subjects & in patients with proven ischemic heart disease.

Methods:

1. Patients will be invited for two endothelial function tests 1 week apart.
2. ECG, heart rate & blood pressure will be recorded at rest prior to each test.
3. Following overnight fasting and discontinuation of all medications for ≥ 12 hours and absence of > 48 hour caffeine consumption, patients will receive 200 mg of caffeine tablets or placebo, in a double-blind, cross-over study design. An hour later the patient will undergo endothelium-dependent flow-mediated dilation (FMD) and endothelium-independent, nitroglycerin (NTG)-mediated vasodilation will be assessed non-invasively in the brachial artery, using a high resolution (15 MHz) linear array ultrasound.
4. Prior to and after the FMD, blood will be drawn to test caffeine levels, adiponectin, CBC, electrolytes, CRP and lipids.

ELIGIBILITY:
Inclusion Criteria:

* Patients with documented ischemic heart disease
* Healthy subjects who are not heavy regular coffee drinkers

Exclusion Criteria:

* Patients with unstable angina pectoris
* Patients with acute or chronic heart failure
* Patients with cardiac arrhythmia

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2007-11; Primary Completion 2009-09 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Flow-mediated dilation (FMD) as surrogate of brachial artery endothelial function | 1-2 hours post caffeine (or placebo)

SECONDARY OUTCOMES:
Markers of inflammation such as hs-CRP, Il6, homocysteine, serum caffeine level | 1-2 hours post caffeine or placebo

CONTACTS AND LOCATIONS:
Overall Officials: Michael Shechter, MD, MA, Principal Investigator — Heart Institute, Chaim Sheba Medical Center, Tel Aviv University; Guy Shalmon, RD, Study Director — Tel Aviv University
Locations (1):
- Heart Institute, Chaim Sheba Medical Center, Tel Litwinsky, Israel